# The Mesh-RTL Project for Prevention of Incisional Hernia. Clinical Trial of Non-inferiority to Compare Two Aponeurotic Closure Techniques in Midline Laparotomy in Patients With Elevated Risk for Hernia.

Sponsor: Hospital Regional de Alta Especialidad del Bajio

Responsible Party: Principal Investigator

Investigator: Edgard Lozada [elozada] Official Title: Master in clinical research

Affiliation: Hospital Regional de Alta Especialidad del Bajio

Collaborators: Juan Carlos Mayagoitia Gonzalez

Eduardo Flores Gonzalez

Approval Number: CI/HRAEB/2018/008

Board Name: Comité de ética en investigación Board Affiliation: CNBCEI-11-CEI-004-20170731

Friday October 18th 2019

#### **Introduction:**

The laparotomy is a surgical incision into the abdomen cavity performed to examine the abdominal and retroperitoneal organs. It is classified according to the medical indication: exploratory, therapeutic, stagemaker, and recently added "damage-control" laparotomy.

There exists so many ways to access the abdominal cavity, usually in relation with the organ or structure to treat; being classified in midline laparotomy, paramedian, transversal, oblique, abdominal-thoracic, etc.

Either an emergency or scheduled procedure, the more usual and functional continues being the midline laparotomy, since it allows a broader and faster approach, with less bleeding and easily to extend if it becomes necessary.

Both the evisceration/eventration and the hernia are considered the most frequent complication of the midline laparotomy with a high morbidity and mortality related. Conditions that will require a second intervention, in Mexico represent the seventh cause of elective surgery and fourth cause of emergency procedures.

So far only the use of the mesh has proven useful in reducing this complication. Our group published in 2016 a clinical trial where it showed that the technique is safe and effective to reduce the presence of incisional hernia, however the use of the mesh brings with it problems such as cost, possibility and use in contaminated cavities and postoperative pain Therefore, the use of the RTL technique as an alternative means to this will help to have one more option for the management of patients with a high risk of incisional hernia.

### **Problem Statement:**

Does the RTL closing technique in the midline laparotomy has the same incident of herniation than the close with supraaponeurotic mesh in patient with elevated risk?

#### Justification

The presence of postincisional hernia need to be considerate as a serious disease, insomuch as it carry on highs rates of morbimortality. The presence of this eventuality is among 0.4-1.2% in elective

surgery and up to 30% in emergency procedures.

It is calculated in de U.S.A. an approximate of 1 million of reinterventions a year to correct this condition, with the respective monetary, time and suffering cost to the patient and the health system.

Given the seriousness, the ultimate global consensus has determinate three main axes to the surgical community to board:

- Identify the relevance of the problem
- Improve the theoretical knowledge and technical capacity in the closing of the abdominal wall
- Implement prophylactic measures in the patients, especially in those with elevated risk.

With the present study we aim to contribute to this global recommendations, comparing two closing techniques of the abdominal wall after a midline laparotomy in patients with elevated risk of herniation. Both techniques are proved safe and useful in other studies, with no comparison to date.

Demonstrate that the use of RTL technique has a similar incidence of herniation than the mesh, in an attempt to prevent postincisional hernias after a midline laparotomy, will bring to the surgical community a cheaper and practical alternative to the mesh.

## **Objectives:**

#### General:

To determinate if the incidence of post-incisional hernia in patients with high risk after a midline laparotomy are similar between the closure of the abdominal wall with the RTL technique and the supraaponeurotic mesh closure reinforcement.

# Specifics:

- To identify the patients with high risk using de validated HERNIA-Project Score.
- To determinate the incidence of post-incisional hernia after one year of the initial midline laparotomy.
- To compare the incidence of post-incisional hernia between the two groups.
- To describe the complications related to each closure technique.

## **Hypothesis:**

## Ho Hypothesis:

There is no difference in the incidence of post-incisional hernia between the RTL technique and the reinforcement with supraaponeurotic mesh closure wall.

## H1 Hypothesis:

There is difference in the incidence of post-incisional hernia between the RTL technique and the reinforcement with suprapponeurotic mesh closure wall.

## Sample size:

The sample size was calculated according to the formula published by Bouemn et all 2015, and based on the results of Kholer and collaborators 2019, where they found in which a percentage of

success was estimated with the standard treatment of 18.5% compared to the experimental management of 7.2%, with a margin of no less than 3%, with an alpha for a tail of 0.05%, and a beta of 20%, with a percentage of estimated losses of approximately 10%, a total of 195 patients per group was obtained.

Statistical analysis Date are presented as frequency and percentage, comparisons between groups were using the  $\chi 2$  test for binary data or Fisher's exact test. Continuous variables are presented as median and range interquartile range and were compared using the Mann-Whitney U-test or t student test if they meet normal criteria. p-Values of less than 0.05 were considered significant. Statistical analyses were performed with SPSS version 25.0.0. Analysis by intention to treat was used.

Study Type: Interventional Primary Purpose: Treatment Study Phase: Phase 4

Interventional Study Model: Parallel Assignment

Clinical trial of non-inferiority

Number of Arms:

Masking: Triple (Participant, Care Provider, Investigator)

Allocation: Randomized
Enrollment: 390 [Anticipated]

## **Primary Outcome Measure**:

#### 1. Incisional Hernia

any abdominal wall gap with or without bulge in the area of a postoperative scar perceptible or palpable by clinical exemination

[Time Frame: 12 and 24 months]

Secondary Outcome Measures:

# 2. postoperative complications

an undesirable and unintended result of an operation affecting the patient that occurs as a direct result of the operation. Haematoma, Facial dehiscence, mesh removal, ileus, reinterventions, re-admissions and death

[Time Frame: 1 month, 1 and 2 years]

## **Elegibility:**

Minimum Age: 18 Years
Maximum Age: 70 Years
Sex: All
Gender Based: No

Accepts Healthy Volunteers: Yes

Criteria:

Inclusion Criteria:

- Patients older than 18 years undergoing midline laparotomy, independently of diagnostic or condition, elective or emergency surgery
- Patients with a score equal or greater than 7 of the hernia score
- Patients who accept to participate and sign the informed consent

#### **Exclusion Criteria:**

- Patients managed with open abdomen or with the impossibility of close the wall
- Patients who had a previous incisional hernia or patients who are participing in anohter trial
- Patients with a life expectative less than 12 months
- Pregnant patients Patients with the antecedent of rejection of prosthesic material

Revised Hernia Score.

```
Revised HERNIAscore = 1 \times (BMI \ge 25 \text{ kg/m}^2) + (1 \text{ COPD}) + (5 \times \text{ extended laparoscopy}) + (6 \times \text{ laparotomy}) + (3 \times \text{ earlier abdominal operation})
```

The revised HERNIAscore was developed and low risk was assigned 0 to 6.9 points, medium risk was assigned 7.0 to 9 points, and high risk was assigned ≥9 points.

#### **Arms and interventions:**

Active Comparator: Onlay Mesh Reinforcement group

The midline fascia was closed with running, slowly absorbable sutures (PDS 1-0) with a recommended suture length to wound length ratio of 4:1. An anterior plane with a width of about 8 cm was created between the anterior fascia and the subcutis. A Lightweight polypropylene mesh was used and placed on the anterior rectus fascia with an overlap of 3 cm. The mesh was fitted in the dissected space and it was fixed with PDS 2-0 suture. Fixing points are placed taking the mesh and the anterior fascia of the rectus muscle, at a distance of 3 cm between each point until completing its circumference.

Experimental: RTL reinforcement group

The RTL suture is placed parallel at a distance of 0.5 cm from the fascial margin. Ideally the thread should lie between the anterior and the posterior rectus muscle sheath; there should be no contact with the rectus muscle. A nonabsorbable monofilamental polypropylene thread and a 65-mm ½ needle are used. Around this longitudinal thread, the continuous suture for fascial closure is introduced immediately lateral to the thread; with running, slowly absorbable sutures (PDS 1-0) with a recommended suture length to wound length ratio of 4:1. An anterior plane with a width of about 8 cm was created between the anterior fascia and the subcutis.



#### References

Medina Ramírez O, Martínez Munive A. Hernias recurrentes y eventración posoperatoria. En: Consejo Mexicano de Cirugía General. Tratado de Cirugía General. Editorial Manual Moderno. México DF. 2009. p. 263-288

Pelissier E, Armstrong O, Ngo P. Anatomía quirúrgica y vías de acceso del abdomen. EMC Elsevier Masson, Paris. 2011; 40-040: 1-40.

Shell DH 4th, de la Torre J, Andrades P, Vasconez LO. Open repair of ventral incisional hernias. Surg Clin North Am. 2008 Feb;88(1):61-83, viii. doi: 10.1016/j.suc.2007.10.008. Review.

PubMed

ID: 18267162

van't RM, De Vos Van Steenwijk PJ, Bonjer HJ, Steyerberg EW, Jeekel J. Incisional hernia after repair of wound dehiscence: incidence and risk factors. Am Surg. 2004 Apr;70(4):281-6.

PubMed

ID: 15098775

Ramirez Barba EJ, Lozano R, Lara Lona E. Epidemiologia de las hernias de la pared abdominal. En: Mayagoitia González JC, hernias de la pared abdominal. Tratamiento actual. 2 ed. Mexico; Editorial Alfil; 2009. p 9-11.

Halm JA, Lip H, Schmitz PI, Jeekel J. Incisional hernia after upper abdominal surgery: a randomised controlled trial of midline versus transverse incision. Hernia. 2009 Jun;13(3):275-80. doi: 10.1007/s10029-008-0469-7. Epub 2009 Mar 4. PubMed ID: 19259615

Le Huu Nho R, Mege D, Ouaïssi M, Sielezneff I, Sastre B. Incidence and prevention of ventral incisional hernia. J Visc Surg. 2012 Oct;149(5 Suppl):e3-14. doi: 10.1016/j.jviscsurg.2012.05.004. Epub 2012 Nov 9. Review. PubMed ID: 23142402

Webster C, Neumayer L, Smout R, Horn S, Daley J, Henderson W, Khuri S; National Veterans Affairs Surgical Quality Improvement Program. Prognostic models of abdominal wound dehiscence after laparotomy. J Surg Res. 2003 Feb;109(2):130-7. PubMed ID: 12643854

van Ramshorst GH, Nieuwenhuizen J, Hop WC, Arends P, Boom J, Jeekel J, Lange JF. Abdominal wound dehiscence in adults: development and validation of a risk model. World J Surg. 2010 Jan;34(1):20-7. doi: 10.1007/s00268-009-0277-y. PubMed ID: 19898894

Gómez CJ, Pere RC. Validación de un modelo de evisceración. Cir Esp. 2013. http://dx.doi.org/10.1016/j.ciresp.2012.12.0088

Goodenough CJ, Ko TC, Kao LS, Nguyen MT, Holihan JL, Alawadi Z, Nguyen DH, Flores JR, Arita NT, Roth JS, Liang MK. Development and validation of a risk stratification score for ventral incisional hernia after abdominal surgery: hernia expectation rates in intra-abdominal surgery (the HERNIA Project). J Am Coll Surg. 2015 Apr;220(4):405-13. doi: 10.1016/j.jamcollsurg.2014.12.027. Epub 2015 Jan 2. PubMed ID: 25690673

Cherla DV, Moses ML, Mueck KM, Hannon C, Ko TC, Kao LS, Liang MK. External Validation of the HERNIAscore: An Observational Study. J Am Coll Surg. 2017 Sep;225(3):428-434. doi: 10.1016/j.jamcollsurg.2017.05.010. Epub 2017 May 26. PubMed ID: 28554782

Marwah S, Marwah N, Singh M, Kapoor A, Karwasra RK. Addition of rectus sheath relaxation incisions to emergency midline laparotomy for peritonitis to prevent fascial dehiscence. World J Surg. 2005 Feb;29(2):235-9. PubMed ID: 15654663

Niggebrugge AH, Trimbos JB, Hermans J, Steup WH, Van De Velde CJ. Influence of abdominal-wound closure technique on complications after surgery: a randomised study. Lancet. 1999 May 8;353(9164):1563-7. PubMed ID: 10334254

Abbott DE, Dumanian GA, Halverson AL. Management of laparotomy wound dehiscence. Am Surg. 2007 Dec;73(12):1224-7. PubMed ID: 18186376

Hollinsky C, Sandberg S. A biomechanical study of the reinforced tension line. A technique for abdominal wall closure and incisional hernias. European surgery. 2007. 39. 2. 122-127

Hollinsky C, Sandberg S. Measurement of the tensile strength of the ventral abdominal wall in comparison with scar tissue. Clin Biomech (Bristol, Avon). 2007 Jan;22(1):88-92. Epub 2006 Aug 10. PubMed ID: 16904247

Hollinsky C, Sandberg S, Kocijan R. Preliminary results with the reinforced tension line: a new technique for patients with ventral abdominal wall hernias. Am J Surg. 2007 Aug;194(2):234-9.

PubMed

ID: 17618812

Lozada-Hernandez EE, Mayagoitia-Gonzalez JC, Smolinski KR, AlvarezCanales JJ, Montiel Hinojosa L, Hernandez Villegas L. Comparacion de dos tecnicas de sutura para

cierre aponeurotico en laparotomia media en pacientes con alto riesgo para evisceracion posquirurgica. Rev Hispanoamericana Hernia.2016; 4(4): 137-143

Bhangu A, Fitzgerald JE, Singh P, Battersby N, Marriott P, Pinkney T. Systematic review and meta-analysis of prophylactic mesh placement for prevention of incisional hernia following midline laparotomy. Hernia. 2013 Aug;17(4):445-55. doi: 10.1007/s10029-013- 1119-2. Epub 2013 May 28. Review. PubMed ID: 23712289

López-Cano M, Pereira JA, Lozoya R, Feliu X, Villalobos R, Navarro S, Arbós MA, Armengol-Carrasco M. PREBIOUS trial: a multicenter randomized controlled trial of PREventive midline laparotomy closure with a BIOabsorbable mesh for the prevention of incisional hernia: rationale and design. Contemp Clin Trials. 2014 Nov;39(2):335-41. doi: 10.1016/j.cct.2014.10.009. Epub 2014 Nov 1. PubMed ID: 25445313

Caro-Tarrago A, Olona Casas C, Jimenez Salido A, Duque Guilera E, Moreno Fernandez F, Vicente Guillen V. Prevention of incisional hernia in midline laparotomy with an onlay mesh: a randomized clinical trial. World J Surg. 2014 Sep;38(9):2223-30. doi: 10.1007/s00268-014-2510-6.

PubMed ID: 24663481

Jairam AP, Timmermans L, Eker HH, Pierik REGJM, van Klaveren D, Steyerberg EW, Timman R, van der Ham AC, Dawson I, Charbon JA, Schuhmacher C, Mihaljevic A, Izbicki JR, Fikatas P, Knebel P, Fortelny RH, Kleinrensink GJ, Lange JF, Jeekel HJ; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement versus primary suture only in midline laparotomies (PRIMA): 2-year follow-up of a multicentre, double-blind, randomised controlled trial. Lancet. 2017 Aug 5;390(10094):567-576. doi: 10.1016/S0140-6736(17)31332-6. Epub 2017 Jun 20. Erratum in: Lancet. 2017 Aug 5;390(10094):554. PubMed ID: 28641875

Bouman AC, ten Cate-Hoek AJ, Ramaekers BL, Joore MA. Sample Size Estimation for Non-Inferiority Trials: Frequentist Approach versus Decision Theory Approach. PLoS One. 2015 Jun 15;10(6):e0130531. doi: 10.1371/journal.pone.0130531. eCollection 2015. PubMed ID: 26076354